CLINICAL TRIAL: NCT02637544
Title: Wirksamkeit Von Akupunktur Auf Den Nicht Chronifizierten Schmerz Bei Craniomandibulärer Dysfunktion - Eine Randomisierte, Placebokontrollierte Klinische Studie
Brief Title: Treatment Efficiency of Acupuncture in Non Chronified Pain Patients With TMDs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Heidelberg Medical Center (Other)
Responsible Party: Principal Investigator, Sinan Sen, Dr. med. dent., University of Heidelberg Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S-099/2014
Record Dates: First submitted 2015-10-01; First posted 2015-12-22 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Temporomandibular Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verum (Active Comparator): Acupuncture therapy.
  For this study arm following acupuncture points suitable for facial pain, according to traditional chinese medicine, were chosen:
  F2, F3, F34, IT3, IT19, S7, T21 and temporomandibular joint ear acupuncture points. Only intervention is the acupuncture therapy.
  Interventions: Other: acupuncture
- Placebo (Placebo Comparator): Placebo acupuncture therapy. For this study arm points outside of the meridians according to traditional chinese medicine, were chosen. Only intervention is the acupuncture therapy.
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — classical acupuncture therapy

SUMMARY:
Aim of this randomized clinical trial is to examine the treatment effectiveness of an acupuncture protocol in adult patients with non chronified TMDs.

DETAILED DESCRIPTION:
Therefore there are two treatment arms, acupuncture verum and acupuncture placebo. Investigators will evaluate for 4 weeks primary current pain, secondary the unassisted jaw opening.

ELIGIBILITY:
Inclusion Criteria:

* non chronified TMD pain
* written informed consent

Exclusion Criteria:

* dysfunctional TMD pain
* systematic diseases affecting the joints or pain perception
* pregnancy
* needle phobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
current pain measured on Numerical Rating Scale | 4 weeks

SECONDARY OUTCOMES:
maximum unassisted jaw opening in mm | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sinan Sen, Dr.med.dent., Principal Investigator — Department of Orthodontics, University of Heidelberg
Locations (1):
- Poliklinik für Hals-Nasen-Ohrenheilkunde, Heidelberg, Germany

REFERENCES:
- [Background] Ezzo J, Berman B, Hadhazy VA, Jadad AR, Lao L, Singh BB. Is acupuncture effective for the treatment of chronic pain? A systematic review. Pain. 2000 Jun;86(3):217-225. doi: 10.1016/S0304-3959(99)00304-8. PMID 10812251
- [Result] Dworkin SF, LeResche L. Research diagnostic criteria for temporomandibular disorders: review, criteria, examinations and specifications, critique. J Craniomandib Disord. 1992 Fall;6(4):301-55. No abstract available. PMID 1298767